CLINICAL TRIAL: NCT02704273
Title: INCEPTUS: A Prospective, Non-Interventional Clinical Assessment Study in X Linked Myotubular Myopathy (XLMTM) Subjects Aged 3 Years and Younger
Brief Title: A Clinical Assessment Study in X-Linked Myotubular Myopathy (XLMTM) Subjects
Acronym: INCEPTUS
Status: Completed | Type: Observational
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: ATX-MTM-009 INCEPTUS
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: X-linked Myotubular Myopathy
Keywords: MTM; XLMTM
MeSH Terms: conditions — Myopathies, Structural, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a pre-Phase 1 prospective, non interventional clinical assessment study to evaluate XLMTM subjects aged 3 years and younger. Many of these clinically relevant measures have not yet been routinely assessed in this population and may provide important insight on the natural history of XLMTM and for future evaluation of potential therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of XLMTM resulting from a confirmed mutation in the MTM1 gene
* Subject is male
* Subject is aged less than 4 years
* Subject requires some mechanical ventilatory support (eg, ranging from 24 hours per day full time mechanical ventilation, to noninvasive support such as continuous positive airway pressure [CPAP] or bilevel positive airway pressure [BiPAP] during sleeping hours)
* Access to subject's medical records
* Signed informed consent by the parent(s) or legally authorized representative(s) (LAR) (when applicable)
* Subject and parent(s) or LAR are willing and able to comply with study visits and study procedures

Exclusion Criteria:

* Subject is participating in an interventional study designed to treat XLMTM
* Subject born <35 weeks gestation who is still not to term as per corrected age
* Subject has a clinically important condition, or life-threatening disease other than XLMTM, in the opinion of the investigator
* Subject has received pyridostigmine or any medication to treat XLMTM within 30 days of enrollment

Max Age: 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: XLMTM subjects aged 3 years and younger.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-07; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Characterize the disease course and natural history of XLMTM using respiratory assessment of strength as measured by PImax | 3 months to 2 years
Characterize the disease course and natural history of XLMTM using neuromuscular assessments, as measured by CHOP INTEND/MFM-20 | 3 months to 2 years

SECONDARY OUTCOMES:
Characterize quality of life as measured by PedsQL | 3 months to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Rico, MD, PhD, Study Director — Audentes Therapeutics
Locations (8):
- United States (4):
  - UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - National Institute of Neurological Disorders and Stroke/NIH Porter, Bethesda, Maryland
- Hospital for Sick Children, Toronto, Ontario, Canada
- Hopital Armand Trousseau, Paris, France
- Ludwig-Maximilians Universität München, Munich, Germany
- Great Ormond Street Hospital, London, United Kingdom